CLINICAL TRIAL: NCT04525846
Title: A Comparison of Urinary Incontinence During Third Trimester of Nulliparous on Pelvic Floor Muscle Training in Rajavithi Hospital
Brief Title: A Comparison of Urinary Incontinence During Third Trimester of Nulliparous on Pelvic Floor Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 072/2562
Record Dates: First submitted 2019-09-10; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; pelvic floor muscle training; nulliparous; pregnancy
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: To compare urinary incontinence, qaulity of life, duration of second stage of labor between pelvic floor muscle training(PFMT) group and nonPFMT group Researcher assess pelvic floor muscle strength by Brink score who verified by urogynecologist , given PFMT program and VDO education, follow up by telephone for compliance, and reassess pelvic floor muscle strength at 4 weeks after consented
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFMT group (Experimental): Researcher was trained and test pelvic floor muscle strength by urogynecologist with Brink scores, participants PFMT group were educated by VDO and recieved program of PFMT after consented form 4 weeks reassess Brink score for check compliance of PFMT and followed up by telephone weekly about compliance of PFMT, general symptom, notice self recording book total 12 weeks and evaluate urinary incontinence by UDI-6 questionaires at third trimester
  Interventions: Other: PFMT
- non PFMT (Experimental): Randomized to non PFMT group watchful waiting until 36-38 week gestation follow up and evaluate UI by UDI6 questionaires at third trimester sames as intervention group
  Interventions: Other: non PFMT

INTERVENTIONS:
Other: PFMT — * program of PFMT consist of contract and hold pelvic floor muscle 10 seconds and relax 10 seconds 20 times per set totally 3 set per day
  * follow up by telephone once a week about compliance of program PFMT, general symptoms, notice recording book
  * at third trimester evaluate UI by questionaire (UDI-6, IIQ-7)
  Arms: PFMT group
Other: non PFMT — Randomized to non PFMT group follow up and evaluate UI at third trimester sames as intervention group
  Arms: non PFMT

SUMMARY:
Comparison of urinary incontinence during third trimester of nulliparous on pelvic floor muscle training in Rajavithi hospital

DETAILED DESCRIPTION:
Outcomes

1. primary outcome >> UI at third trimester
2. secondary outcome >> quality of life, duration of second stage of labor

   * Inclusion criteria nulliparous GA 20-24 week gestation singleton Age 18-35 years old Can communicate and understand Thai language Cooperating to join research
   * Exclusion criteria DFIU Maternal medical condition or high risk pregnancy such as multifetal gestation, chronic hypertension, pregestational DM, epilepsy, autoimmune disease, polyhydramnios asthma
   * Pre-excisting urinary incontinence
   * prepregnancy BMI>=30 kg/m2
   * smoking
   * 2 groups study >> control and intervention group
   * Both groups were evaluated urinary incontinence(UI) at third trimester with UDI-6 and IIQ-7 questionaires
   * Intervention group was trianed pelvic floor muscle strength and evaluate strength with Brink score by researcher who was trained and tested pelvic floor muscle strength by urogynecologist at day 1 then reassess Brink score at 4 weeks
   * program of pelvic floor muscle training ( PFMT) consist of contract and whole pelvic floor muscle 10 seconds and relaxation 10 second total 20 times per set total 3 set per day
   * intervention group was followed up once a week by telephone about compliance of program, general symptom and notice for self recording sheet
   * PFMT program follow up total 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* nulliparous
* gestational gae 20-24 week
* age 18-35 year
* can communicate and understand Thai language
* co-operate to join research

Exclusion Criteria:

* DFIU
* maternal medical condition or high risk pregnancy such as multifetal gestation , pregestational DM, chonic hypertension , epilepsy, autoimmune disease, polyhydramnios, asthma
* pre-excisting urinary incontinence
* prepregnant BMI >=30 kg/m2
* smoking

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 150 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence at third trimester both group | GA 36-38 wk
  Use Questionaires Urinary Distress Inventory (UDI-6) include 6 domains( Frequency, Urgency incontinence, Stress incontinence, Drops, Emptying difficulty, Pain /discomfort each domain raw score from 0-3 (0=not at all, 1= a little bit, 2=moderately, 3=greatly) (total raw score 18 point ) define score total 100 point if at least 16.7% means urinary incontinence and below 16.7% means nornal ( continence= no UI )

SECONDARY OUTCOMES:
Quality of life at third trimester both group | GA 36-38 wk
  Incontinence impact questionaires (IIQ-7) includes Household chores, Physical recreation, Entertainment activities, Travel ability, Social activities, Emotional health, Feeling frustrated. Each domain has raw score 0-3 (0=not at all, 1= a little bit, 2=moderately, 3=greatly), total raw score 21 points. It's defined total score 100 point if at least 70 means impact qaulity of life
Duration of second stage of labor in both group | date of delivery
  use partograph and labor record, Duration of second stage of labor define as times of cervical fully dilatation until baby delivery difine as minutes
Correlation between urinary incontinence and quality of life | GA 36-38 wk
  questionaire UDI-6 , IIQ-7 hypothesis high score of UDI6 associated poor quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rogers RG, Ninivaggio C, Gallagher K, Borders AN, Qualls C, Leeman LM. Pelvic floor symptoms and quality of life changes during first pregnancy: a prospective cohort study. Int Urogynecol J. 2017 Nov;28(11):1701-1707. doi: 10.1007/s00192-017-3330-7. Epub 2017 Apr 17. PMID 28417155
- [Result] ICS. A Background to urinary and faecal incontinence. August 2015
- [Result] Bekele A, Adefris M, Demeke S. Urinary incontinence among pregnant women, following antenatal care at University of Gondar Hospital, North West Ethiopia. BMC Pregnancy Childbirth. 2016 Oct 28;16(1):333. doi: 10.1186/s12884-016-1126-2. PMID 27793178
- [Result] Tanawattanacharoen S, Thongtawee S. Prevalence of urinary incontinence during the late third trimester and three months postpartum period in King Chulalongkorn Memorial Hospital. J Med Assoc Thai. 2013 Feb;96(2):144-9. PMID 23936978
- [Result] Niamhom S. Nursing process in caring for postpartum mothers with stress urinary incontinence. J Nurs Sci. 2009; 27(1): 22-31
- [Result] Zhu L, Li L, Lang JH, Xu T. Prevalence and risk factors for peri- and postpartum urinary incontinence in primiparous women in China: a prospective longitudinal study. Int Urogynecol J. 2012 May;23(5):563-72. doi: 10.1007/s00192-011-1640-8. Epub 2012 Jan 26. PMID 22278711
- [Result] Sangsawang B, Sangsawang N. Is a 6-week supervised pelvic floor muscle exercise program effective in preventing stress urinary incontinence in late pregnancy in primigravid women?: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2016 Feb;197:103-10. doi: 10.1016/j.ejogrb.2015.11.039. Epub 2015 Dec 2. PMID 26720598
- [Result] สรวีร์ วีระโสภณ, อภิรักษ์ สันติงามกุล. การทดสอบความแม่นยำของแบบสอบถามประเมินภาวะกลั้นปัสสาวะไม่ได้ (IIQ-7 UDI-6) เมื่อแปลเป็นภาษาไทย. จุฬาลงกรณ์เวชสาร 2559; 60(4): 389-98
- [Result] Kok G, Seven M, Guvenc G, Akyuz A. Urinary Incontinence in Pregnant Women: Prevalence, Associated Factors, and Its Effects on Health-Related Quality of Life. J Wound Ostomy Continence Nurs. 2016 Sep-Oct;43(5):511-6. doi: 10.1097/WON.0000000000000262. PMID 27607747
- [Result] Sangsawang B, Sangsawang N. Stress urinary incontinence in pregnant women: a review of prevalence, pathophysiology, and treatment. Int Urogynecol J. 2013 Jun;24(6):901-12. doi: 10.1007/s00192-013-2061-7. Epub 2013 Feb 23. PMID 23436035
- [Result] Okunola TO, Olubiyi OA, Omoya S, Rosiji B, Ajenifuja KO. Prevalence and risk factors for urinary incontinence in pregnancy in Ikere-Ekiti, Nigeria. Neurourol Urodyn. 2018 Nov;37(8):2710-2716. doi: 10.1002/nau.23726. Epub 2018 Jun 8. PMID 29882369
- [Result] Schreiner L, Crivelatti I, de Oliveira JM, Nygaard CC, Dos Santos TG. Systematic review of pelvic floor interventions during pregnancy. Int J Gynaecol Obstet. 2018 Oct;143(1):10-18. doi: 10.1002/ijgo.12513. Epub 2018 May 18. PMID 29705985
- [Result] Lin YH, Chang SD, Hsieh WC, Chang YL, Chueh HY, Chao AS, Liang CC. Persistent stress urinary incontinence during pregnancy and one year after delivery; its prevalence, risk factors and impact on quality of life in Taiwanese women: An observational cohort study. Taiwan J Obstet Gynecol. 2018 Jun;57(3):340-345. doi: 10.1016/j.tjog.2018.04.003. PMID 29880161
- [Result] Pelaez M, Gonzalez-Cerron S, Montejo R, Barakat R. Pelvic floor muscle training included in a pregnancy exercise program is effective in primary prevention of urinary incontinence: a randomized controlled trial. Neurourol Urodyn. 2014 Jan;33(1):67-71. doi: 10.1002/nau.22381. Epub 2013 Feb 6. PMID 23389863
- [Result] Kahyaoglu Sut H, Balkanli Kaplan P. Effect of pelvic floor muscle exercise on pelvic floor muscle activity and voiding functions during pregnancy and the postpartum period. Neurourol Urodyn. 2016 Mar;35(3):417-22. doi: 10.1002/nau.22728. Epub 2015 Feb 3. PMID 25648223
- [Result] Salvesen KA, Stafne SN, Eggebo TM, Morkved S. Does regular exercise in pregnancy influence duration of labor? A secondary analysis of a randomized controlled trial. Acta Obstet Gynecol Scand. 2014 Jan;93(1):73-9. doi: 10.1111/aogs.12260. Epub 2013 Nov 7. PMID 24102423
- [Result] Morkved S, Bo K, Schei B, Salvesen KA. Pelvic floor muscle training during pregnancy to prevent urinary incontinence: a single-blind randomized controlled trial. Obstet Gynecol. 2003 Feb;101(2):313-9. doi: 10.1016/s0029-7844(02)02711-4. PMID 12576255
- [Result] Hundley AF, Wu JM, Visco AG. A comparison of perineometer to brink score for assessment of pelvic floor muscle strength. Am J Obstet Gynecol. 2005 May;192(5):1583-91. doi: 10.1016/j.ajog.2004.11.015. PMID 15902162
- [Result] Botros S, Gandhi S, Abramov Y, Sand P, Nickolov A, Goldberg R. Normotive values for the short forms of the UDI and IIQ in community dwelling women.